CLINICAL TRIAL: NCT02374931
Title: Pilot Investigation of 18F-FES PET/CT Imaging of Desmoid Tumors
Brief Title: 18F-FES PET/CT in Imaging Patients With Desmoid Tumors
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ashish Patel, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC SAR 1458; NCI-2015-00081 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICC SAR 1458 (Other: Vanderbilt-Ingram Cancer Center); P30CA068485 (NIH)
Record Dates: First submitted 2015-02-16; First posted 2015-03-02 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Deep Fibromatosis/Desmoid Tumor; Familial Adenomatous Polyposis
Keywords: desmoid; FES-PET; aggressive fibromatosis
MeSH Terms: conditions — Desmoid Tumors; Adenomatous Polyposis Coli | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (18F-FES PET/CT) (Experimental): Patients undergo 18F-FES PET/CT imaging over 30 minutes.
  Interventions: Drug: F-18 16 Alpha-Fluoroestradiol; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: F-18 16 Alpha-Fluoroestradiol — Undergo 18F-FES PET/CT
  Other Names: 16 alpha-fluroestradiol-17 beta; F-18 FES; FES; Fluorine-18 16 alpha-fluoroestradiol
Procedure: Positron Emission Tomography — Undergo 18F-FES PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan
Procedure: Computed Tomography — Undergo 18F-FES PET/CT
  Other Names: CAT; CAT Scan; CT
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies fluorine (F)-18 16 alpha-fluoroestradiol (18F-FES) positron emission tomography (PET)/computed tomography (CT) in imaging patients with desmoid tumors. 18F-FES binds to estrogen receptors, which are present on desmoid tumors, and gives off radiation that may be detected by PET and CT scans. The PET/CT scan forms an image that may show where tumor cells with estrogen receptors can be found in the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the avidity of desmoid tumors on 18F-FES PET/CT imaging. II. Correlate 18F-FES PET avidity with degree of estrogen receptor (ER) expression by immunohistochemistry (IHC).

OUTLINE:

Patients undergo 18F-FES PET/CT imaging over 30 minutes.

After completion of study, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven extra-abdominal desmoid tumors
* Not currently on estrogen medication for birth control, menopause, or other reason
* No anti-estrogen therapy for desmoid tumor within the past 6 months
* Both sporadic desmoid tumors and those associated with familial adenomatous polyposis (FAP) syndromes will be included

Exclusion Criteria:

* Pregnancy or nursing patients
* Patients who do not wish to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-04; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Standard uptake value (SUV) measured as percent injected dose per cc | Initial visit, average within 24 hours of imaging
  Data will be summarized graphically and numerically. Continuous variables (e.g. SUV) will be summarized using the mean, standard deviation, and a 5 number percentile summary set (minimum, p25, p50, p75, and maximum). The Spearman correlation statistic will be used to estimate the magnitude of a linear association between SUV and IHC measures. Ninety-five percent confidence intervals will be calculated for all point estimates.

SECONDARY OUTCOMES:
IHC staining intensity in tissue samples | Within 4 weeks of imaging done at initial visit, day 1
  IHC staining intensity measured on an ordinal scale or dichotomized as positive or negative. Data will be summarized graphically and numerically. Categorical measures (e.g., IHC) will be summarized in frequency tables. The Spearman correlation statistic will be used to estimate the magnitude of a linear association between SUV and IHC measures. Ninety-five percent confidence intervals will be calculated for all point estimates.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Patel, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://vicc.org/ct/